CLINICAL TRIAL: NCT07283211
Title: Using a NAO Robot to Enhance Occupational Therapy for Children With Cerebral Palsy
Brief Title: NAO Robot in Pediatric Occupational Therapy
Acronym: NAO Robot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Medipol University (Other)
Collaborators: Medipol University (Other); Yeditepe University (Other)
Responsible Party: Principal Investigator, Hilal Bostancı Seçkin, LECTURER, Ankara Medipol University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: E-10840098-772.02-30; 123E355 (Other Grant/Funding Number: The Scientific and Technological Research Council of Turkey (TUBITAK 1002))
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-11

CONDITIONS: Cerebral Palsy (CP); Activities of Daily Living
Keywords: occupational therapy; cerebral palsy; social robots
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Group - Occupational Therapy With and Without Social Robot Support (Experimental): This single-group arm includes all participants, who receive two sequential phases of occupational therapy. In Phase 1, children receive routine occupational therapy sessions delivered by a licensed occupational therapist. After a 2-week interval, participants enter Phase 2, during which they receive the same occupational therapy activities supplemented with robot-assisted interaction using the NAO humanoid robot. All participants experience both phases in the same order, and no randomization or group allocation is performed.
  Interventions: Other: Occupational Therapy Intervention; Other: NAO Robot-Assisted Occupational Therapy

INTERVENTIONS:
Other: Occupational Therapy Intervention — Routine Occupational Therapy. Participants receive standard occupational therapy sessions delivered by a licensed pediatric occupational therapist. Sessions include individualized therapeutic activities targeting fine motor skills, bilateral coordination, sensory processing, activities of daily living (ADL) training, and play-based functional tasks.
Other: NAO Robot-Assisted Occupational Therapy — NAO Robot-Assisted Occupational Therapy. Participants receive the same core occupational therapy program as in Phase 1, supplemented with robot-mediated interaction using the NAO humanoid robot (SoftBank Robotics).

SUMMARY:
Cerebral Palsy (CP) is a non-progressive neurological disorder that affects movement and posture, often impairing upper extremity function and daily activity performance. Technological tools, such as social robots, have shown promise in supporting rehabilitation. This study investigated the effects of NAO robot-assisted therapy on functional performance, motivation, and emotional states in children with unilateral CP.

Sixteen children participated in a 14-week intervention, which included 12 weeks of task-oriented therapy. In six of those weeks, sessions incorporated the NAO robot, which simulated three daily activities identified using the Canadian Occupational Performance Measure (COPM) and offered motivational feedback. Emotional responses were tracked using the Empatica E4 wristband, measuring blood volume pulse (BVP), electrodermal activity (EDA), and skin temperature (ST).

DETAILED DESCRIPTION:
This single-group interventional study investigated the effect of adding the social humanoid robot NAO to occupational therapy sessions on upper extremity function, hand skills, and motivation in children with unilateral spastic cerebral palsy (CP). Sixteen children aged 5-15 years, classified as GMFCS I-III, MACS 1-3, CFCS 1-2, and MAS 0-2, participated.

The study consisted of two sequential 6-week phases:

Phase 1: Routine occupational therapy sessions (40 minutes each).

Phase 2: Routine occupational therapy supplemented with NAO robot-assisted activities (same duration).

Sessions targeted functional tasks identified using the Canadian Occupational Performance Measure (COPM), such as eating, throwing a ball, and brushing teeth. Upper extremity function was assessed with the Quality of Upper Extremity Skills Test (QUEST); functional abilities with PEDI; activity limitations and bimanual hand use with GMFCS and BFMF; and occupational performance and satisfaction with COPM.

Physiological signals (blood volume pulse, electrodermal activity, and skin temperature) were recorded using the Empatica E4 wristband to assess children's motivation and emotional responses during sessions. Data were analyzed using appropriate statistical methods, including t-tests, Mann-Whitney U, Friedman test, and Wilcoxon signed-rank tests with Bonferroni correction.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5-15 years
* Diagnosis of unilateral spastic cerebral palsy
* Classified as Level I-III according to the Gross Motor Function Classification System (GMFCS)
* Classified as Level 1-3 on the Manual Ability Classification System (MACS)
* Level 0-2 on the Modified Ashworth Scale, indicating mild to moderate spasticity

Exclusion Criteria:

* History of upper extremity orthopedic surgery within the past year
* Presence of epileptic symptoms
* Receipt of botulinum toxin treatment within the last six months

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2025-06-02 (Actual)

PRIMARY OUTCOMES:
Quality of Upper Extremity Skills Test (QUEST) | 20 minutes
Pediatric Evaluation of Disability Inventory (PEDI) | 10 minutes
Bimanual Fine Motor Function | 10 minutes
Canadian Occupational Performance Measure | 10 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Medipol University, Altindağ, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Due to the inclusion of pediatric participants and the sensitive nature of the clinical data, individual participant data will not be shared.